CLINICAL TRIAL: NCT06540612
Title: Effects of Aerobic Exercise on Cancer-Related Biomarkers, Functional Capacity, Cognitive Status and Quality of Life in Women With Breast Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Nahide Fidancioglu, PhD Student, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TABED 1-24-82
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Female; Quality of Life; Survivorship
Keywords: Breast Cancer; Rehabilitation; Biomarkers; Exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise Intervention (Experimental): In this group, participants do moderate-intensity aerobic exercise three days a week.
  Interventions: Other: Aerobic exercise
- Physical activity counseling (Active Comparator): Realistic and achievable goals are set based on the individual's needs and goals. An individualized exercise program is created. This program may include aerobic exercise, strength training, flexibility exercises, and other activities. The individual is educated about proper techniques, safe practices, and benefits of the exercises. The individual's progress is monitored and evaluated regularly, and adjustments to the program are made as needed. Ongoing support and encouragement is provided to help the individual stay motivated and achieve their goals.
  Interventions: Behavioral: Physical activity counseling
- control group (No Intervention): The control group continued their current daily activities and did not perform any new exercise program.

INTERVENTIONS:
Other: Aerobic exercise — Aerobic exercise is a set of physical activities that work large muscle groups continuously and rhythmically.
  Arms: Aerobic Exercise Intervention
Behavioral: Physical activity counseling — Physical activity counselling is a service that provides personalized guidance and support to help individuals adopt a healthy lifestyle.
  Arms: Physical activity counseling

SUMMARY:
This study aims to emphasize the exercise-induced changes in some circulating biomarkers (CRP, IGF-1(insulin like growth factor), insulin, leptin, IL-6(interleukin-6) , TNF-α(tumor necrosis factor), adiponectin), quality of life, functional capacity, cognitive functions and after aerobic exercise in women diagnosed with breast cancer in remission period.

The women who will participate in the study consist of breast cancer survivors aged 18-65 years.

The hypothesis of this study:

Exercise program in women diagnosed with breast cancer in remission positively affects the levels of circulating biomarkers CRP, IGF-1, insulin, leptin, IL-6, TNFα and adiponectin, and improves quality of life, functional capacity, and cognitive functions.

Participants will be divided into 3 groups. The first group will receive moderate intensity aerobic exercise 3 times a week for 12 weeks. The second group will receive physical activity counseling by a physiotherapist for 12 weeks. The third group will continue their daily routines and no intervention will be performed. The evaluations will be repeated three times for all three groups: at baseline, after six weeks and after twelve weeks.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumor in women with a rate of 30%. Again, 15% of cancer-related deaths in women are due to breast cancer. Breast cancer, whose incidence among women is increasing in our country, is seen in one out of every four women diagnosed with cancer. Approximately one in every eight women is at lifelong risk of developing breast cancer (Turkish Society of Medical Oncology Breast Cancer, 2019).

As a side effect of the disease and multimodal anticancer interventions, breast cancer patients may experience cancer-related physical and psychological symptoms such as cancer-related fatigue, decreased muscle mass, loss of strength, decreased functional capacity, and pain. These symptoms create a vicious cycle leading to deterioration in quality of life. Oncological rehabilitation aims to reduce such symptoms through multimodal, transprofessionally delivered, goal-oriented and person-centered coordinated interventions. Oncological rehabilitation is available before, during, between and after cancer treatments.

Inflammation is the hallmark of cancer and is associated with poor clinical outcomes in patients with various types of solid tumors. Inflammation activates certain signaling pathways to promote cell survival, proliferation, migration and invasion. Preclinical studies show that reducing inflammation and targeting inflammatory signaling pathways slows cell growth and delays tumor progression. Furthermore, obesity causes chronic inflammation that can promote malignant cell growth. The anti-inflammatory benefit of aerobic exercise may arise in part due to a reduction in adiposity.

Decreased immune function often accompanies anti-cancer therapies and reduces overall quality of life. Compromised chronic inflammation and cellular immunity are major concerns, as both promote a pro-tumor environment that may contribute to disease progression. Therefore, there is a need to identify options to manage inflammation while maximizing immune function in cancer survivorship. Exercise is a potentially attractive option. However, the role of exercise training on immune function and inflammatory markers is not well addressed in current exercise oncology guidelines.

Immune cell rates and function provide direct evidence of immunity in cancer survivors. Cytokines are often categorized as pro- or anti-inflammatory; some function as both (such as interleukin-6). Higher circulating levels of pro-inflammatory cytokines are linked to cancer-related outcomes. For example, breast cancer patients with advanced tumors have higher circulating levels of tumor necrosis factor (TNF) compared with healthy individuals. Previous systematic reviews had concluded that exercise training had no effect on circulating cytokines in cancer survivors overall. However, a recent meta-analysis using a more homogeneous population reported positive effects of TNF, interleukin-6, interleukin-8 and interleukin-2 in breast cancer. Despite the role of the inflammatory state in various cancers and the growing body of literature examining cytokines in exercise oncology, it remains unclear whether the benefits of exercise extend beyond breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65
* Literate
* Diagnosed with stage 2 breast cancer
* Completed primary breast cancer treatment at least 6 months ago (excluding hormone therapy/aromatase inhibitors)
* Provided cooperation
* Female
* Patients who are willing and willing to participate in the study

Exclusion Criteria:

* Those who are using psychotic, anxiolytic, antidepressant, analgesic and sleeping pills
* Those with metastasis
* Those with a history of lymphedema
* Those with neurological disease
* Those who are pregnant or breastfeeding
* Uncontrolled hypertensive patients
* Those who are incapable of verbal communication or physical movement

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 69 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Quality Of Life Questionnaire | A total of three assessments will be made at the beginning of the study, at the end of 6 weeks, and at the end of 12 weeks.
  Developed by the European Organization for Research and Treatment of Cancer, it is a multidimensional quality of life scale. This scale developed by Aaronson et al. consists of 30 questions in total. It consists of three subscales: 1-The Functional Scale consists of physical, role, cognitiv, emotional and social subscales. 2-General Health Statuse; 3-Symptom Scale consists, fatigue, nausea, vomiting, pain, shortness of breath, sleep disturbance, loss of appetite, constipation , diarrhea , and financial impact. The 28 questions on the functional and symptom scales consist of four options for each question: not at all (1 point), a little (2 points), quite a bit (3 points), a lot (4 points). In the general health scale, there are options from 1 to 7 points ranging from very poor to excellent. The lowest total score that patients can get from the functional score, symptom score and general health score is 0 and the highest score is 100.

SECONDARY OUTCOMES:
Functional Capacity | A total of three assessments will be made at the beginning of the study, at the end of 6 weeks, and at the end of 12 weeks.
  The six-minute walk test for the assessment of functional capacity will be performed according to the American Thoracic Society criteria. The six-minute walk test will be performed on a flat, unobstructed surface. Heart rate, blood pressure, oxygen saturation, dyspnea and fatigue levels according to the modified Borg scale will be determined before and after the test. The content of the test will be explained to the participants. During the test, the participants will be told that they will walk at their daily walking pace for 6 minutes and that they can stop and rest whenever they want. All participants will be tested to walk for 6 minutes and their walking distances will be measured and recorded. The test will be repeated 2 times at 20 minute intervals. In the measurements, all protocols applied in the first test will be applied again. The first results will be used for patients who do not participate in the retest.

OTHER OUTCOMES:
Cognitive Status | A total of three assessments will be made at the beginning of the study, at the end of 6 weeks, and at the end of 12 weeks.
  The Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) Questionnaire will be used to assess the cognitive status of individuals. FACT-COG is a form filled out by the patient to assess chemotherapy-induced behavioral cognitive impairment and treatment, questioning the last 7 days. This form, evaluates cognitive sensitivity, attention and coordination, memory, verbal fluency, functional interference, observations of others about the individual, change in functionality compared to before and quality of life parameters. It consists of 4 sub-headings: The questions in the sections of perceived cognitive impairments, other people's comments, perceived cognitive skills and impact on quality of life are scored between 0-4. The perceived cognitive impairments and perceived cognitive abilities subsections contain the opposite questions and the last 2 questions are not included in the scoring. Increasing total score indicates improving cognitive function.
Biomarkers(CRP, IGF-1, insulin, leptin, IL-6, TNF-α, adiponectin) | A total of three assessments will be made at the beginning of the study, at the end of 6 weeks, and at the end of 12 weeks.
  After an eight-hour overnight fast, venous blood samples will be collected from the antecubital vein in a sitting position. Dry tubes (BD Vacutainer, SST II Advance, Austria) with gel separator containing clot activator will be used for serum collection. Blood samples will be centrifuged at 3500 rpm for 10 min and serum will be separated. Sera will be stored in a deep freezer (Nüve DF 290, Turkey) at -80˚C. Starting from the day before the day of analysis, the frozen samples will be gradually thawed at -20˚C, +4˚C and room temperature, respectively. In order to avoid repeated freezing and thawing, laboratory work will be performed after all samples have been collected. Standards, kits and sera will be brought to room temperature (18- 26°C). Serum samples will be analyzed according to routine laboratory procedures. All parameters will be run in 2 replicates.

CONTACTS AND LOCATIONS:
Overall Officials: Nahide Fidancıoğlu, Principal Investigator
Locations (1):
- Nahide FIDANCIOGLU, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Result] Asher A, Myers JS. The effect of cancer treatment on cognitive function. Clin Adv Hematol Oncol. 2015 Jul;13(7):441-50. PMID 26353040
- [Result] Erratum: ATS Statement: Guidelines for the Six-Minute Walk Test. Am J Respir Crit Care Med. 2016 May 15;193(10):1185. doi: 10.1164/rccm.19310erratum. No abstract available. PMID 27174486
- [Result] Aggarwal BB, Gehlot P. Inflammation and cancer: how friendly is the relationship for cancer patients? Curr Opin Pharmacol. 2009 Aug;9(4):351-69. doi: 10.1016/j.coph.2009.06.020. Epub 2009 Aug 6. PMID 19665429
- [Result] Furman D, Campisi J, Verdin E, Carrera-Bastos P, Targ S, Franceschi C, Ferrucci L, Gilroy DW, Fasano A, Miller GW, Miller AH, Mantovani A, Weyand CM, Barzilai N, Goronzy JJ, Rando TA, Effros RB, Lucia A, Kleinstreuer N, Slavich GM. Chronic inflammation in the etiology of disease across the life span. Nat Med. 2019 Dec;25(12):1822-1832. doi: 10.1038/s41591-019-0675-0. Epub 2019 Dec 5. PMID 31806905
- [Result] Iyengar NM, Gucalp A, Dannenberg AJ, Hudis CA. Obesity and Cancer Mechanisms: Tumor Microenvironment and Inflammation. J Clin Oncol. 2016 Dec 10;34(35):4270-4276. doi: 10.1200/JCO.2016.67.4283. Epub 2016 Nov 7. PMID 27903155
- [Result] Bower JE, Greendale G, Crosswell AD, Garet D, Sternlieb B, Ganz PA, Irwin MR, Olmstead R, Arevalo J, Cole SW. Yoga reduces inflammatory signaling in fatigued breast cancer survivors: a randomized controlled trial. Psychoneuroendocrinology. 2014 May;43:20-9. doi: 10.1016/j.psyneuen.2014.01.019. Epub 2014 Jan 30. PMID 24703167
- [Result] Johnson DE, O'Keefe RA, Grandis JR. Targeting the IL-6/JAK/STAT3 signalling axis in cancer. Nat Rev Clin Oncol. 2018 Apr;15(4):234-248. doi: 10.1038/nrclinonc.2018.8. Epub 2018 Feb 6. PMID 29405201
- [Result] Zomkowski K, Wittkopf PG, Baungarten Hugen Back B, Bergmann A, Dias M, Sperandio FF. Pain characteristics and quality of life of breast cancer survivors that return and do not return to work: an exploratory cross-sectional study. Disabil Rehabil. 2021 Dec;43(26):3821-3826. doi: 10.1080/09638288.2020.1759150. Epub 2020 May 12. PMID 32393077
- [Result] Khosravi N, Stoner L, Farajivafa V, Hanson ED. Exercise training, circulating cytokine levels and immune function in cancer survivors: A meta-analysis. Brain Behav Immun. 2019 Oct;81:92-104. doi: 10.1016/j.bbi.2019.08.187. Epub 2019 Aug 24. PMID 31454519
- [Result] Kokkonen K, Saarto T, Makinen T, Pohjola L, Kautio H, Jarvenpaa S, Puustjarvi-Sunabacka K. The functional capacity and quality of life of women with advanced breast cancer. Breast Cancer. 2017 Jan;24(1):128-136. doi: 10.1007/s12282-016-0687-2. Epub 2016 Mar 22. PMID 27002988
- [Result] Al Maqbali M, Al Sinani M, Al Naamani Z, Al Badi K, Tanash MI. Prevalence of Fatigue in Patients With Cancer: A Systematic Review and Meta-Analysis. J Pain Symptom Manage. 2021 Jan;61(1):167-189.e14. doi: 10.1016/j.jpainsymman.2020.07.037. Epub 2020 Aug 5. PMID 32768552
- [Result] Mantovani A, Allavena P, Sica A, Balkwill F. Cancer-related inflammation. Nature. 2008 Jul 24;454(7203):436-44. doi: 10.1038/nature07205. PMID 18650914
- [Result] Klassen O, Schmidt ME, Ulrich CM, Schneeweiss A, Potthoff K, Steindorf K, Wiskemann J. Muscle strength in breast cancer patients receiving different treatment regimes. J Cachexia Sarcopenia Muscle. 2017 Apr;8(2):305-316. doi: 10.1002/jcsm.12165. Epub 2016 Nov 28. PMID 27896952
- See also: EORTC QLQ-C30 Scoring Manual — http://www.eortc.org/app/uploads/sites/2/2018/02/SCmanual.pdf
- See also: Breast Cancer — http://www.kanser.org/saglik/toplum/kanser-turleri-alt-kategori/meme-kanseri